CLINICAL TRIAL: NCT04806386
Title: The Role of Fiber in the Prevention and Treatment of Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kyle Staller, MD, MPH, Assistant Professor in Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000691
Record Dates: First submitted 2021-03-08; First posted 2021-03-19 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-11

CONDITIONS: Fecal Incontinence; Irritable Bowel Syndrome With Diarrhea
Keywords: IBS-D; IBS; FI; Fecal Incontinence; Irritable Bowel Syndrome with Diarrhea; Irritable Bowel Syndrome
MeSH Terms: conditions — Fecal Incontinence; Irritable Bowel Syndrome | interventions — Psyllium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Psyllium fiber supplement treatment (Experimental): All patients will receive psyllium fiber in the form of edible bars, 7g, twice a day to total 14g per day.
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Dietary Supplement: Psyllium — Psyllium fiber powder baked into a bar is commonly used as a first line of treatment for patients with fecal incontinence.

SUMMARY:
The purpose of this study is to determine the effect of fiber supplementation on the fecal metagenome and metabolome in relation to symptoms and anorectal physiology in post-menopausal women with irritable bowel syndrome with diarrhea suffering from liquid stool fecal incontinence (FI.)

DETAILED DESCRIPTION:
This is an open-label, single-arm study at Massachusetts General Hospital that aims to recruit post-menopausal female patients with solid stool fecal incontinence. The investigators hope that subjects taking a daily fiber supplement will experience reduced episodes and symptoms of fecal incontinence, measured through quality of life questionnaires and daily stool and food diaries. Subjects will undergo 2 anorectal manometry procedures. Stool samples will also be collected for metabolomic and metagenomic analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Female, post-menopausal
2. Age 50-90 years old
3. BMI >18.5 and <40 kg/m2
4. Rome IV criteria for liquid stool fecal incontinence occurring at least twice per month
5. At least one FI episode during the run-in period
6. Compliant with reporting during run-in (completion of two 3-day food diaries and two 7-day bowel diaries)
7. Submission of two stool samples during the run-in period
8. Ability to follow verbal and written instructions
9. Informed consent form signed by the subjects

Exclusion Criteria:

1. Less than two episodes per month of liquid stool fecal incontinence
2. Non-compliance with reporting during run-in
3. Patients reporting laxative, enema, and/or suppository usage during the run-in period
4. GI tract structural abnormality that would increase likelihood of obstruction
5. Dysphagia, swallowing disorder, or history of esophageal structural lesions
6. History of GI lumen surgery within 60 days prior to entry into the study
7. Neurological disorders, metabolic disorders, or other significant disease that would impair their ability to participate in the study
8. Inability to tolerate or contraindication to performance of anorectal manometry
9. Celiac disease, Crohn's disease, ulcerative colitis
10. Current anorectal fistula and/or abscess
11. Age <50 or >90
12. BMI of <18.5 or ≥40 kg/m2
13. History of allergic reaction to psyllium
14. Previous trial of soluble fiber supplementation for fecal incontinence within the previous 30 days
15. History of sacral nerve stimulator or artificial anal sphincter placement
16. Administration of investigational products within 1 month prior to Screening Visit
17. Subjects anticipating surgical intervention during the study

19. History of intestinal stricture (e.g., Crohn's disease) 20. History of intestinal obstruction or subjects at high risk of intestinal obstruction including suspected small bowel adhesions 21. History of malabsorption 22. Any other clinically significant disease interfering with the assessments of psyllium, according to the Investigator (e.g., disease requiring corrective treatment, potentially leading to study discontinuation) 23. Any relevant biochemical abnormality interfering with the assessments of psyllium, according to the Investigator 24. Patients with metallic implants within a 30 cm radius of the TAMS electromagnetic coil 25. Currently on opioids 26. Patients with severe cardiac disease, chronic renal failure, or previous GI surgery EXCEPT cholecystectomy, appendectomy, Nissen fundoplication, and partial colectomy 27. Patients with neurological diseases and increased intracranial pressure 28. Patients with impaired cognizance 29. Previous pelvic surgery/radiation, radical hysterectomy 30. Patients with Ulcerative Colitis or Crohn's Disease 31. History of or current rectal prolapse 32. Previous history of anal fissure, anal surgery (abscess), congenital anorectal malformation, fistulae or inflamed hemorrhoids 33. Pregnant women 34. Use of antibiotics in previous 60 days

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Stool metagenomics | Change from baseline to final visit. Through study completion, up to 6 weeks.
  Sequence-based microbial community surveys will be carried out to characterize rare taxa and understand relationships between community membership and function from stool samples collected from baseline to the final visit.
Stool microbiome | Change from baseline to final visit. Through study completion, up to 6 weeks.
  Stool samples will be shipped to Metabolon Inc, for metabolomics profiling on a well-validated high-throughput metabolomics platform. Sample prep and global metabolomics profiling will be conducted using four liquid chromatography tandem mass spectrometry methods that measure four complementary sets of metabolite classes. Metabolite peaks are quantified using area-under-the curve. Raw area counts for each metabolite in each sample are normalized to correct for variation resulting from inter-day tuning differences by setting the medians to 1.0 for each run. Metabolites are identified by automated comparison of the ion features in the experimental samples to a reference library of ~8,000 chemical standard entries that are curated for quality control using Metabolon software. Coefficients of variations (CVs) will be measured in blinded quality control samples randomly distributed among study samples, and we will analyze and control for batch variation.

SECONDARY OUTCOMES:
Fecal incontinence severity index (FISI) | Change from baseline to final visit. Through study completion, up to 6 weeks.
  Questionnaire about the severity of symptoms in those with fecal incontinence. Consists of 4 questions, each rated on a scale of 1 to 6. Lower scores indicate higher severity of symptoms. (Min, 4, max 24)
Fecal Incontinence quality of life (FIQL) | Change from baseline to final visit. Through study completion, up to 6 weeks.
  Questionnaire about the quality of life of those with fecal incontinence. Questions are rated from 1 to 4 in each section. Lower rating represent worse quality of life. Subscales exist for lifestyle, coping behavior, embarrassment, and depression. There is no total score for this outcome, only subscores per section. (Min 4, max, 16)
Anorectal manometry parameters | Change from baseline to final visit. Through study completion, up to 6 weeks.
  Anorectal manometry (ARM) procedure performed to measure the change in anal and rectal muscle function and sensation at baseline and at the final visit.
Translumbosacral anorectal magnetic stimulation | Change from baseline to final visit. Through study completion, up to 6 weeks.
  Translumbosacral anorectal magnetic stimulation (TAMS) performed during the ARM procedure to measure the change in the nerve conduction between the spinal cord and rectum at baseline and at the final visit.
Global assessment of relief | Change from baseline to final visit. Through study completion, up to 6 weeks.
  A 7-point scale indicating overall fecal incontinence symptom relief where 1 represents completely relieved and 7 represents completely worse.
Bloating scale | Change from baseline to final visit. Through study completion, up to 6 weeks.
  A 10-point scale indicating bloating severity where 0 represents the least severity and 10 represents the most severity
Urgency scale | Change from baseline to final visit. Through study completion, up to 6 weeks.
  A 10-point scale indicating urgency severity where 0 represents the least severity and 10 represents the most severity
Flatus scale | Change from baseline to final visit. Through study completion, up to 6 weeks.
  A 10-point scale indicating flatus severity where 0 represents the least severity and 10 represents the most severity
Waist circumference measurement (cm) | Change from baseline to final visit. Through study completion, up to 6 weeks.
  A measure of the subject's waist circumference in the area where the most bloating is experienced

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Staller, MD MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No